CLINICAL TRIAL: NCT06436469
Title: Mindfulness-based Stress Reduction Programs to Reduce Compassion Fatigue in Nurses
Brief Title: MBSR Programs to Reduce Compassion Fatigue in Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Ruthlande Nore, Principal Investigator, Nova Southeastern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-280-NSU
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Compassion Fatigue
MeSH Terms: conditions — Compassion Fatigue | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: The model for this study is a single-group pretest-posttest design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness interventions (Other): The intervention involves participation in a structured Mindfulness-Based Stress Reduction (MBSR) program. Participants engage in a series of sessions over a four week period. During these sessions, participants learn and practice mindfulness techniques such as deep breathing and body scans.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR) Program

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) Program — The intervention involves participation in a structured Mindfulness-Based Stress Reduction (MBSR) program. Participants engage in a series of sessions over a four week period. During these sessions, participants learn and practice mindfulness techniques such as deep breathing and body scans. The program is designed to enhance participants' awareness of their thoughts, emotions, and bodily sensations in the present moment, promoting a nonjudgmental acceptance of their experiences. By cultivating mindfulness skills, participants aim to reduce stress, enhance emotional regulation, and develop resilience in coping with the challenges of their work environment.

SUMMARY:
The goal of this observational study is to evaluate the effectiveness of a mindfulness-based stress reduction (MBSR) program in reducing compassion fatigue among nurses. The main question it aims to answer is:

Does participation in an MBSR program decrease levels of compassion fatigue among nurses? The primary hypothesis is that nurses who participate in the MBSR program will experience a significant reduction in compassion fatigue after implementing the interventions.

Participants will include psychiatric nurse practitioners working in high-stress environments.

Participants will:

Attend a series of MBSR sessions over a specified period. Engage in mindfulness practices such as body scans, and deep breathing. Complete self-report measures to assess levels of compassion fatigue before and after the intervention.

DETAILED DESCRIPTION:
This observational study aims to assess the impact of a mindfulness-based stress reduction (MBSR) program on reducing compassion fatigue among psychiatric nurse practitioners working in high-stress environments. The primary question it seeks to address is whether participation in the MBSR program leads to decreased levels of compassion fatigue among nurses.

The primary hypothesis posits that nurses who engage in the MBSR program will experience a significant reduction in compassion fatigue following the intervention.

Participants in this study will be psychiatric nurse practitioners who work in demanding healthcare settings. These individuals will be invited to participate voluntarily in the MBSR program.

The intervention will involve participants attending a series of MBSR sessions conducted over a specified period, typically lasting around 4 weeks. During these sessions, participants will be guided through various mindfulness practices, including body scans and deep breathing exercises. These techniques are designed to enhance participants' awareness of their thoughts, emotions, and bodily sensations, promoting a nonjudgmental acceptance of their experiences.

To assess the effectiveness of the intervention, participants will complete self-report measures to evaluate their levels of compassion fatigue. These assessments will be administered both before the start of the MBSR program (baseline/pretest) and after its completion (follow-up/posttest). By comparing pre- and post-intervention scores, researchers will evaluate any changes in compassion fatigue levels among participants.

Overall, this study aims to contribute to our understanding of the potential benefits of mindfulness-based interventions in mitigating compassion fatigue among psychiatric nurse practitioners, with implications for improving the well-being and resilience of healthcare professionals in high-stress environments.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric Nurse Practitioner
* At least one year of nursing experience
* Participants would need to be able to read and understand English.

Exclusion Criteria:

* Is not a Psychiatric Nurse practitioner
* Reservations against the program
* Have <1 yr. nursing experience

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-11 (Actual); Study Completion 2024-08-11 (Actual)

PRIMARY OUTCOMES:
Compassion Fatigue Assessment | Participants will complete the compassion fatigue assessment at two time points: before starting the mindfulness-based stress reduction (MBSR) program (baseline/pretest) and after completing the program (follow-up/posttest) over a period of 4 weeks.
  The primary outcome measure involves assessing participants' levels of compassion fatigue using a validated instrument, such as the Professional Quality of Life (ProQOL) questionnaire. This questionnaire evaluates various dimensions of compassion fatigue, including emotional exhaustion, depersonalization, and reduced personal accomplishment.

CONTACTS AND LOCATIONS:
Overall Officials: Charmaine Coffman, Study Chair — Nova Southeastern University
Locations (1):
- My Psychiatrist, Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The IPD sharing plan involves sharing anonymized participant data (demographics, baseline characteristics, outcome measures, intervention details) for collaboration, further analysis, or meta-analyses. Before sharing, informed consent will be obtained, and identifying information will be removed to protect confidentiality. Sharing will comply with institutional policies, ethical guidelines, and data sharing agreements, ensuring regulatory and privacy compliance.
Supporting Information: SAP
Time Frame: The data from this observational study will become available for sharing after completion of the study and publication of the primary study findings and will be available for up to 36 months after.
Access Criteria: Access criteria for obtaining anonymized IPD include: clear research purpose related to compassion fatigue, affiliation with recognized institutions, ethical approval evidence, compliance with data security protocols, signing data sharing agreements, and adherence to regulatory requirements.